CLINICAL TRIAL: NCT02922270
Title: Outcome and Risk Factors For Mortality in Peritoneal Dialysis Patients: 20 Years Experience in a Single Turkish Center
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Director, Istanbul University
Other Study IDs: 252
Record Dates: First submitted 2016-09-19; First posted 2016-10-04 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Therapeutic Procedural Complication
Keywords: peritoneal dialysis: outcome; peritoneal dialysis: complications; peritoneal dialysis: technique; peritoneal dialysis: peritonitis
MeSH Terms: interventions — Risk Factors; Mortality

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Who have received PD as renal replacement therapy (RRT) over a period of 20 years.
  Interventions: Other: Peritoneal dialysis patients at the Istanbul Medical Faculty

INTERVENTIONS:
Other: Peritoneal dialysis patients at the Istanbul Medical Faculty — The aims of this study were to evaluate patient and technique survival rates, investigate peritonitis rates and evaluate factors affecting mortality in peritoneal dialysis (PD) patients over a period of 20 years at Istanbul Faculty of Medicine Peritoneal Dialysis Unit.
  Other Names: OUTCOME AND RISK FACTORS FOR MORTALITY

SUMMARY:
INTRODUCTION AND AIMS: The aims of this study were to evaluate patient and technique survival rates, investigate peritonitis rates and evaluate factors affecting mortality in peritoneal dialysis (PD) patients over a period of 20 years at Istanbul Faculty of Medicine Peritoneal Dialysis Unit.

METHODS: Two hundred seventy seven patients have received PD as renal replacement therapy (RRT) over a period of 20 years. After exclusion of patients with follow-up shorter than 3 months and patients whose data were not available, 250 patients were examined retrospectively. Data for sex, age, primary disease, comorbidities, follow up duration, cause of death, and cause of technique failure were collected from medical records.

DETAILED DESCRIPTION:
Material and Method All patients 18 years of age and older who were treated with PD at the Istanbul Medical Faculty from October 1994 to October 2014 were included in the study. Patients exclude which follow-up shorter than 3 months and patients whose data were not available. From the day PD was started, all peritonitis data were collected prospectively in a large database. The data include Socio-demographic data, type of peritoneal dialysis, starting time and duration of every peritonitis episode, causative organisms and outcome of the peritonitis, which could be cure, change of PD catheter, transfer to hemodialysis, or death. The time in months from PD start to the first episode of peritonitis was computed.

Primary kidney disease was classified into 9 main categories according to the codes of the European Renal Association - European Dialysis and Transplant Association. Peritonitis in PD was defined as a peritoneal dialysate effluent containing >100 white blood cells/mL, of which >50% were polymorphonuclear leukocytes. Patients with two or more pathogens isolated from the cultures in a peritonitis episode were considered to have polymicrobial peritonitis. A relapse of peritonitis was defined when the same organism or a culture-negative peritonitis episode was identified within 4 weeks of completing appropriate antibiotic therapy for a previous episode.

Socio-demographic, clinical and treatment characteristics, medium (standard deviation for continuous variables) or median (25th and 75th percentages); number for categorical variables (rate) were calculated. Cox regression analysis applied to examine the impact of demographic and clinical features of periton dialysis patients . Chi-square test for categorical variables used. Univariate and multivariate analyzes calculated using the Kruskal-Wallis or Mann-Whitney test method. P-value was <0.05 for as long as it is considered statistically significant. The evaluation of the results obtained using SPSS 21.0 software.

ELIGIBILITY:
Inclusion Criteria:

* all patients 18 years of age and older
* treated with PD at the Istanbul Medical Faculty from October 1994 to October 2014

Exclusion Criteria:

* follow-up shorter than 3 months and patients whose data were not available,
* data were not available
* patients who were unwilling
* patients who unable to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred seventy seven patients have received PD as renal replacement therapy (RRT) over a period of 20 years.
Sampling Method: Probability Sample
Enrollment: 277 (Actual)
Dates: Start 1995-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Patient survival | 5 - 10 years

SECONDARY OUTCOMES:
Treatment failure | 5 - 10 years
  Re-initiation of hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, Dr., Study Chair — Division of Nephrology, Department of Internal Medicine, Istanbul Faculty of Medicine, Istanbul University

IPD SHARING:
Plan to Share IPD: No